CLINICAL TRIAL: NCT03677570
Title: The Relationship Between Postural Stability, Performance and Trunk Muscle Endurance in Female Athletes
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Cagatay Gokdogan, research assisstant, Gazi University
Other Study IDs: CAGATAY1
Record Dates: First submitted 2018-09-18; First posted 2018-09-19 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Sports Physical Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Female athletes: A total of 45 female athletes (15 volleyball, 15 handball, and 15 football players) (average age: 22,26 ± 6,43 / BMI: 21,45 ± 2,39) participated in the study.Trunk muscle endurance of the participants was measured with the McGill core endurance tests and the prone bridge test. Postural stability of the participants was evaluated using Biodex Biosway Portable Balance System (950- 460 USA) device. Sportive performance was tested with the vertical jump test and the hexagonal obstacle test.
  Interventions: Diagnostic Test: postural stability
- Healthy Control: 15 sedentary females (average age: 24,86 ± 3,02 / BMI: 21,42 ± 1,90) participated in the study.Trunk muscle endurance of the participants was measured with the McGill core endurance tests and the prone bridge test. Postural stability of the participants was evaluated using Biodex Biosway Portable Balance System (950- 460 USA) device. Sportive performance was tested with the vertical jump test and the hexagonal obstacle test.
  Interventions: Diagnostic Test: postural stability

INTERVENTIONS:
Diagnostic Test: postural stability — Postural Stability, vertical jump test, hexagonal obstacle test, trunk flexion test, trunk extension test, side bridge test,prone bridge test

SUMMARY:
As core stability improves in handball players, ball-throwing speed increases as well. Postural stability is considered as the most important component of athletic performance as it occurs in almost all movement types. No studies have yet evaluated postural stability, performance and trunk muscle endurance in female athletes at the same time and examined the relationship between these parameters.This study aims to identify the relationship between the postural stability, performance and trunk muscle endurance of female athletes in different branches of sports.

DETAILED DESCRIPTION:
A total of 45 female athletes (15 volleyball, 15 handball, and 15 football players) (average age: 22,26 ± 6,43 / BMI: 21,45 ± 2,39) and 15 sedentary females (average age: 24,86 ± 3,02 / BMI: 21,42 ± 1,90) participated in the study. Trunk muscle endurance of the participants was measured with the McGill core endurance tests and the prone bridge test. Postural stability of the participants was evaluated using Biodex Biosway Portable Balance System (950- 460 USA) device. Sportive performance was tested with the vertical jump test and the hexagonal obstacle test.

ELIGIBILITY:
Inclusion Criteria:

* Not being injured in the last 3 months
* Being a professional athlete that does training 5 days a week for the last two years

Exclusion Criteria:

* cardiovascular system diseases
* pregnant women were excluded

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 45 female athletes and 15 healthy sedentary controls volunteered to take part in the study.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-11-06 (Actual); Primary Completion 2016-01-16 (Actual); Study Completion 2017-01-23 (Actual)

PRIMARY OUTCOMES:
postural stability | Baseline assessment, no follow-up
  stability index
vertical jump test | Baseline assessment, no follow-up
  centimetre
hexagonal obstacle test | Baseline assessment, no follow-up
  second
trunk flexion test | Baseline assessment, no follow-up
  second
trunk extension test | Baseline assessment, no follow-up
  second
prone bride test | Baseline assessment, no follow-up
  second
side bridge test | Baseline assessment, no follow-up
  second

CONTACTS AND LOCATIONS:
Overall Officials: nevin güzel, prof.dr, Study Chair — Faculty of Health Sciences, Department of Physical Therapy and Rehabilitation, Gazi University

IPD SHARING:
Plan to Share IPD: No